CLINICAL TRIAL: NCT06680141
Title: The Effect of Virtual Reality Glasses Used Before Cesarean Section on Surgical Fear and Anxiety
Brief Title: The Effect of Virtual Reality Glasses Used Before Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Director, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/260
Record Dates: First submitted 2024-10-20; First posted 2024-11-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Glasses (Experimental): Among the women who have been admitted for a planned caesarean section, the Informed Consent Form and the Data Collection Form including Sociodemographic Characteristics, Surgical Fear Scale, Spielberg State-Trait Anxiety Scale will be applied to the women who meet the criteria and randomization will be applied. After randomization, they will be divided into a virtual reality glasses application group and a control group. All women will be applied the Spielberg State-Trait Anxiety Scale and Surgical Fear Scale in the patient room before and after the SGG application. The experimental group will be shown a video (30 minutes) of the 9-month fetal development process, with glasses on before going to surgery.
  Interventions: Other: Virtual reality glasses
- control (No Intervention): Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention will perform

INTERVENTIONS:
Other: Virtual reality glasses — control group
  Other Names: control group
  Arms: Virtual Reality Glasses

SUMMARY:
The aim of this study is to determine the effect of Virtual Reality Glasses Used Before Cesarean Section on Surgical Fear and Anxiety

DETAILED DESCRIPTION:
Hypotheses 01; there was no difference between the Surgical Fear and Anxiety score of the Virtual Reality Glasses group and the control group.

The study will be carried out in two different groups. The practice will start with meeting the women whom will go to cesarean section in the hospital. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Virtual Reality Glasses Group; the intervention will be given glasses before the surgery and will be shown a video (30 minutes) of the 9-month fetal development process. Among the women who were admitted for a planned caesarean section, those who met the criteria would first be given the Informed Consent Form and a data collection form including sociodemographic characteristics, surgical fear scale, Spielberg State-Trait Anxiety Scale, and then randomization would be applied.

control group; the first surgical fear scale, anxiety scores will be recorded. After cesarean section anxiety scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo a cesarean section for the first time,
* Are over the age of 18,
* Have no diagnosed mental illness,
* Have no diagnosed physical illness in themselves or their baby,
* Volunteer to participate in the study

Exclusion Criteria:

* Have previously undergone a cesarean section,
* Are under the age of 18,
* Have a diagnosed mental illness,
* Have a diagnosed physical illness in themselves or their baby, Do not volunteer to participate in the study. -

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Spielberger State Anxiety Scale | 30 minutes
  The inventory was developed by Spielberger, Gorsuch, and Lushene in 1970. An adaptation, validity, and reliability study of the State-Trait Anxiety Scale in Turkish was conducted by Oner and Le Compte in 1983. The scale consists of two subdimensions: the state anxiety has 20 items and is used to determine what is felt at a specific moment under certain conditions, and the trait anxiety has 20 items and is used to determine what has been felt in the last 7 days. High scores from each subscale indicate a high level of anxiety. The Cronbach's a for the STAI ranges from 0.83 to 0.87. It will be applied half an hour before the surgery.
Surgical Fear Scale (SFS): | 30 minutes
  The scale was developed by Theunissen et al. (2014) and its validity and reliability for use in Turkey were established by Bağdigen and Karaman Özlü (2018). The scale consists of 8 items in an 11-point Likert format, scored between 0 and 10. It is divided into two subscales, each containing 4 items, measuring short-term and long-term fears related to surgery.
  Items 1-4 assess fear regarding short-term outcomes of surgery, while items 5-8 evaluate fear concerning long-term outcomes. Each item is rated from "0: not afraid at all" to "10: extremely afraid." A higher total score, with a maximum of 26 points, indicates a greater level of fear. In the validity and reliability study, the Cronbach's alpha coefficient for the total score was found to be 0.93.It will be applied half an hour before the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Emine KOÇ, Asst.Prof, Study Chair — Ondokuz Mayıs University; Nazlı Baltacı, Asst.Prof, Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)